CLINICAL TRIAL: NCT04325178
Title: Mycoprotein as the Basis of a Sustainable Diet to Support Muscle Mass Maintenance and Reconditioning in Older Adults.
Acronym: MASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: uexeter
Record Dates: First submitted 2020-03-04; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Aging; Sarcopenia
Keywords: Ageing; Muscle protein synthesis; Resistance exercise; Sarcopenia; Sustainable protein
MeSH Terms: conditions — Sarcopenia | interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal (Experimental): Participants receive the majority of their protein from animal-derived protein sources (1.8g.kg.day).
  Interventions: Other: Protein, calorie and macronutrient controlled diet, derived from either omnivorous or non-animal sources, alongside unilateral resistance exercise, over a three-day period.
- Non-animal (Experimental): Participants receive all their protein from non-animal-derived protein sources (1.8g.kg.day).
  Interventions: Other: Protein, calorie and macronutrient controlled diet, derived from either omnivorous or non-animal sources, alongside unilateral resistance exercise, over a three-day period.

INTERVENTIONS:
Other: Protein, calorie and macronutrient controlled diet, derived from either omnivorous or non-animal sources, alongside unilateral resistance exercise, over a three-day period. — Participants received a control diet either derived from omnivorous or non-animal food sources, providing 1.8g.kg.day of protein, for a three-day period. Calories were calculated and set to place participants in a state of energy balance. Participants completed three bouts of unilateral resistance exercise, 5 sets of 30 maximal concentric knee extension contractions, on each morning that they received the control diet. During this three-day period participants also consumed a deuterium oxide tracer allowing for the measurement of muscle protein synthesis, in rested and exercised tissue, with incremental biopsies.

SUMMARY:
A hallmark of ageing is loss of skeletal muscle mass and strength (sarcopenia). Sarcopenia is explained, partially, by reduced responsiveness of muscle to dietary protein. This 'anabolic resistance' can be overcome by consuming protein in close proximity to exercise and/or adequate amounts across the day. Consequently, there is momentum for a greater protein RDA for older individuals. Concurrently, there is a need to establish an evidence base for the efficacy of non-animal proteins.

Mycoprotein is a sustainable non-animal derived protein that imposes a significantly lower environmental burden than animal sources. Our previous work suggests that mycoprotein has the potential to support muscle tissue remodelling to a similar extent as animal derived protein sources. The study will employ a deuterium oxide tracer to quantify muscle protein synthesis over a period of three days in response to a vegan diet or animal based diet, alongside daily unilateral resistance exercise in older adults.

DETAILED DESCRIPTION:
Dietary protein plays a critical role in the daily regulation of muscle mass by virtue of its ability to regularly stimulate muscle protein synthesis rates. Sarcopenia is mechanistically explained, at least in part, by the reduced responsiveness of older adult's muscle tissue to these anabolic properties of dietary protein. However, this 'anabolic resistance' can be overcome by paying attention to the synergy that exists between the anabolic effects of dietary protein and physical activity. Specifically, consuming dietary protein in close temporal proximity to physical activity and/or adequate amounts of dietary protein per meal is an effective strategy to optimise muscle protein metabolism in older adults. These mechanistic, physiological findings are supported by longitudinal studies showing that older individuals who consume modestly greater amounts of dietary protein than the current RDA, and/or maintain/adopt an active lifestyle, experience reduced rates of sarcopenia and typically live healthier lives.

With the importance of dietary protein to support active, healthy ageing evident, and a consequent scientific momentum moving towards a considerable (≥50%) rise in recommended protein intake for older individuals, the inevitable question arises: 'where should this dietary protein to support healthy ageing come from?' Current and future generations are required to view developments in human nutrition through the lens of mounting challenges associated with the sustainability of increased production of animal proteins, a concern also of primary importance to Quorn Foods. However, research into the nutritional physiology of alternative, sustainable, non-animal derived protein sources is in its infancy, particularly so in older adults. Therefore, there is considerable scientific interest, public health value and commercial opportunity in establishing a robust evidence base for the efficacy of non-animal, sustainably produced dietary protein sources to support active, healthy ageing.

Mycoprotein, a food source produced by continuous fermentation of the filamentous fungus Fusarium venenatum, imposes a significantly lower environmental burden during its production compared with animal sources. In collaboration with Quorn Foods, we recently reported that acute consumption of mycoprotein in young adults results in equivalent amino acid bioavailability to that of milk protein, and therefore shows promise as a protein source to support muscle anabolism and metabolic health in numerous populations. In the present proposal, we wish to translate and extend these findings into the older adult population. We will exploit a stable isotope tracer approach (oral administration of deuterium oxide ['heavy water']) to make in vivo measurements of cumulative, free living muscle protein synthesis rates in response to a highly sustainable, non-animal derived, mycoprotein based diet with or without physical activity, compared with a more traditional diet reliant on animal derived protein sources (matched for total protein). The study will increase our knowledge of how effective non-animal derived proteins are at supporting muscle tissue remodelling in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30
* Recreationally active

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes) (as this may affect normal protein metabolism).
* Any diagnosed cardiovascular disease or hypertension.
* Elevated blood pressure at the time of screening. (An average systolic blood pressure reading of ≥150mmHg over two or more measurements and an average diastolic blood pressure of ≥90mmHg over two or more measurements.)
* Chronic use of statins or diabetic medication.
* A personal or family history of epilepsy, seizures or schizophrenia.
* Allergic to mycoprotein / Quorn, penicillin, or milk.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | Three days.
  Calculation of muscle protein synthesis using the product-precursor method, with deuterium in the body water pool utilised as the precursor and the incorporation of deuterated alanine into muscle tissue as the product.

SECONDARY OUTCOMES:
Resistance-type exercise work done | Three days.
  The work done (J) over 5 sets of 30 isokinetic knee extension contractions, on three consecutive days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No